CLINICAL TRIAL: NCT00102102
Title: PET Evaluation of NK1 Receptor Using [18F]SPA-RQ in Post-Traumatic Stress Disorder
Brief Title: Role of Substance P in Post-Traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050080; 05-M-0080
Record Dates: First submitted 2005-01-20; First posted 2005-01-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Substance P; Neurokinin; Tachykinin; Anxiety; Neuroreceptor Imaging; Post-Traumatic Stress Disorder; PTSD; Healthy Volunteer; HV
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — (2-fluoromethoxy-5-(5-trifluoromethyltetrazol-1-yl)benzyl)(2-phenylpiperidin-3-yl)amine

INTERVENTIONS:
Drug: [18F]SPA-RQ

SUMMARY:
This study will examine the role of substance P, a chemical messenger in the brain, in post-traumatic stress disorder (PTSD), a chronic anxiety disorder. PTSD can develop after exposure to a terrifying event or ordeal, such as a violent personal assault, natural or human-caused disaster, accident, or military combat. Substance P is a peptide that may be important in the response to certain psychiatric and neurological diseases and conditions, including anxiety.

Healthy normal volunteers and people with PTSD who are between 18 and 65 years of age may be eligible for this study. Candidates are screened with a physical examination, blood and urine tests, pregnancy test for women who can become pregnant, and a neuropsychological evaluation.

Participants undergo positron emission tomography (PET) and magnetic resonance imaging (MRI) scanning. An optional lumbar puncture (spinal tap) is also requested.

PET Scanning

PET uses small amounts of a radioactive chemical called a tracer that "labels" active areas of the brain. The tracer used in this study is [18F]SPA-RQ. For the procedure, the subject lies still on the scanner bed. A special mask is fitted to the head to help keep the subject's head still during the scan so the images will be clear. A 20-minute "transmission" scan is done before the radioactive tracer is injected to provide measures of the brain that will help in the precise calculation of information from subsequent scans. After the tracer is injected through a needle in the arm, pictures are taken continuously for about 2 hours. Then, 20- to 40-minute images are taken every hour until about 5 hours after the injection.

MRI Scanning

An MRI scan is scheduled at some time within 1 year of the PET scan. MRI uses a magnetic field and radio waves to obtain images of body tissues and organs. The subject lies still on a table inside the tunnel-like MRI scanner. Earplugs are worn to muffle loud noises that occur during the scanning. The maximum duration of the scan is 60 minutes.

Lumbar Puncture

Lumbar puncture is used to examine the cerebrospinal fluid (CSF) that surrounds both the brain and the spinal cord. For this procedure, a local anesthetic is given to numb the skin in the lower back area. A small needle is then inserted into the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle.

Blood Draw

A blood sample is collected to generate cell lines that can be used to extract DNA (genetic material) for gene studies and that can be frozen for future use.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a chronic, debilitating disorder that places a significant burden on individuals and society. Abnormalities in the serotonergic and noradrenergic systems and dysregulation of the hypothalamic-pituitary adrenal (HPA) axis have been proposed as neurobiological mechanisms in the development of the disorder, however the exact underpinnings of the neurobiology of the disorder must be elucidated.

Distribution of substance P (SP) and its receptor, neurokinin 1 (NK1) receptor, includes regions implicated in the pathophysiology of PTSD, namely the amygdala, hippocampus, hypothalamus, and locus ceruleus. There is a considerable spatial (and therefore functional) overlap between the SP-NK1 receptor system and other neurotransmitter (e.g., norepinephrine, serotonin) pathways with well established roles in anxiety. Preclinical studies indicate that stress regulates levels of SP in several brain regions. In addition, in several animal models, NK1 receptor antagonists demonstrate anxiolytic-like property. These anxiolytic-like effects seem to involve different mechanisms than those of currently available anxiolytics.

In this protocol, we will use a PET ligand that acts as an NK1 receptor antagonist, [18F]SPA-RQ ([18F]-labeled Substance P Antagonist Receptor Quantifier). Using this tracer, we will look for regional differences in NK1 receptor binding in 20 patients with PTSD and 20 healthy controls. The goal of the present study is to demonstrate the involvement of SP in PTSD, and thereby, further our understanding of its role in the psychopathology of this illness.

ELIGIBILITY:
INCLUSION CRITERIA:

PTSD Samples:

Twenty subjects (age 18-65) with current PTSD, as defined by DSM-IV criteria, of any ethnicity without other significant medical conditions will be selected.

Healthy Control Samples:

Twenty healthy subjects (age 18-65) without a known personal or family history of psychiatric disorders in first-degree relatives will be selected.

A control subject will be matched to each subject with PTSD for age, gender, and handedness, respectively.

They must not be actively using illicit drugs or engaged in heavy consumption of alcohol, had no metallic implants that are ferromagnetic, and competent to sign consent forms to participate in the study.

EXCLUSION CRITERIA:

Patients must not have taken antidepressant or other medications likely to alter SP-NK1 receptor system. Effective medications will not be discontinued for the purpose of this study.

Subjects will be excluded if they have:

1. DSM-IV Axis I diagnostic criteria other than PTSD and Major depression (All controls must not meet any of the Axis I diagnoses);
2. DSM-IV criteria for psychoactive substance abuse/dependence within six months;
3. take psychotropic medication in last 3 weeks (8 weeks for fluoxetine);
4. abnormal MRI other than minor atrophy;
5. abnormal laboratory test, including HIV test;
6. are currently pregnant or breast feeding (as documented by pregnancy testing at screening or at days of the scanning);
7. prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits (A total effective dose 5.0 rem in a year and a 5 rad per year to the lens of the eyes, gonads and blood-forming organs; and 15 rad annually for all other organs);
8. are unable to lay on one's back for PET/MRI scans (PET and MRI scans take approximately 5 and 1 hour, respectively);
9. any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.);
10. individuals who recently donated blood;
11. serious suicidal ideation or behavior;
12. Xylocaine allergy;
13. positive HIV test.

For healthy subjects, exclusion criteria b) through m) are same to those for PTSD subjects. As for item a), subjects will be excluded if they meet any current DSM-IV Axis I diagnostic criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Breslau N, Kessler RC, Chilcoat HD, Schultz LR, Davis GC, Andreski P. Trauma and posttraumatic stress disorder in the community: the 1996 Detroit Area Survey of Trauma. Arch Gen Psychiatry. 1998 Jul;55(7):626-32. doi: 10.1001/archpsyc.55.7.626. PMID 9672053
- [Background] Davidson JR, Hughes D, Blazer DG, George LK. Post-traumatic stress disorder in the community: an epidemiological study. Psychol Med. 1991 Aug;21(3):713-21. doi: 10.1017/s0033291700022352. PMID 1946860
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257